CLINICAL TRIAL: NCT06569121
Title: Efficacy of an Evidence-based Telehealth-delivered Weight-loss Intervention to Enhance Access and Reach Underserved Groups After Stroke
Brief Title: Efficacy of a Telehealth Delivered Group Lifestyle Balance for People Post Stroke (tGLB-CVA)
Acronym: tGLB-CVA
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Baylor Research Institute (Other)
Collaborators: National Institute on Disability, Independent Living, and Rehabilitation Research (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: BSW IRB# 024-414
Record Dates: First submitted 2024-08-20; First posted 2024-08-23 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2025-01

CONDITIONS: Stroke, Acute; Stroke; Stroke, Cardiovascular; Stroke (CVA) or TIA; Stroke/Brain Attack
MeSH Terms: conditions — Stroke; Myocardial Infarction

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Wait List Control (WLC) (No Intervention): Participants randomized to the wait list control (WLC) will begin the telehealth Group Lifestyle Balance for People post stroke (tGLB-CVA) intervention 6 months after enrolling into the study and completing a baseline assessment.
- Telehealth Group LIfestyle Balance for People with Stroke (tGLB-CVA) (Experimental): The telehealth Group Lifestyle Balance for People post stroke (tGLB-CVA) is a one-year program with 22 sessions. The tGLB-CVA is a modification of the Diabetes Prevention Program Group Lifestyle Balance (DPP-GLB) developed by the University of Pittsburgh Diabetes Prevention Support Center (DPSC). It begins with 12 weekly sessions called the Core Program, followed by a Transition phase consisting of 2 bi-weekly and 2 monthly sessions, and a Support Phase consisting of 6 monthly sessions. The goal of the tGLB-CVA program is to help the participant achieve and maintain a 5-7% weight-loss through healthy eating and physical activity.
  Interventions: Behavioral: Group Lifestyle Balance for People Post Stroke (GLB-CVA)

INTERVENTIONS:
Behavioral: Group Lifestyle Balance for People Post Stroke (GLB-CVA) — 12-month healthy lifestyle and weight loss program modified from the Diabetes Prevention Program Group Lifestyle Balance (DPP-GLB)
  Arms: Telehealth Group LIfestyle Balance for People with Stroke (tGLB-CVA)

SUMMARY:
Investigators will conduct a randomized controlled trial (RCT) to assess intervention efficacy of telehealth delivery of the GLB-CVA (tGLB-CVA) compared to a 6-month wait-list control (WLC) in partnership with a diverse group of patient partners and peer mentors.

ELIGIBILITY:
Inclusion Criteria:

* Body Mass Index ≥25
* All types of stroke
* Able to Participate in Physical Activity
* ≥12 months post first stroke
* Have internet, phone, or computer access, or be willing to use one provided by the study team

Exclusion Criteria:

* Contraindications for physical activity
* Low Cognitive Function
* Residing in hospital, acute rehab, skilled nursing facility
* Not fluent in the English language
* Pre-existing eating disorder
* Pregnancy

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 94 (Estimated)
Dates: Start 2024-12-07 (Actual); Primary Completion 2027-08-31 (Estimated); Study Completion 2029-12-31 (Estimated)

PRIMARY OUTCOMES:
Body Weight | Baseline, 3, 6, 9, 12, 18 month
  Body weight (lbs) will be captured via self-weighing using provided BodyTrace Smart Scale, which includes cellular connectivity so weight will be sent directly to the research team. The scales have demonstrated good concordance rates with self-weighing in previous research. Scales will be setup by the research team before being mailed to participants with instructions.

SECONDARY OUTCOMES:
Circumference | Baseline, 3, 6, 9, 12, 18 month
  Waist and hip circumference (centimeters) will be collected from a local Quest Diagnostics
Height | Baseline, 3, 6, 9, 12, 18 month
  Height (inches) will be collected from a local Quest Diagnostics
Body Mass Index (BMI) | Baseline, 3, 6, 9, 12, 18 month
  Body Mass Index (BMI, kg/m^2) will be calculated from height and weight from a local Quest Diagnostics
Blood pressure | Baseline, 3, 6, 9, 12, 18 month
  Blood Pressure (mmHg, diastolic and systolic) will be collected at a local Quest Diagnostics
Blood Sugar, Hemoglobin A1c (HbA1c) | Baseline, 3, 6, 9, 12, 18 month
  Fasting venous sample will be obtained for Hemoglobin A1c (HbA1c) at a local Quest Diagnostics and recorded as a parentage.
Blood Glucose | Baseline, 3, 6, 9, 12, 18 month
  Fasting venous sample will be obtained for blood glucose (mg/dL) at a local Quest Diagnostics.
High Density Lipoprotein (HDL) cholesterol | Baseline, 3, 6, 9, 12, 18 month
  Fasting venous sample will be obtained for High Density Lipoprotein (HDL, mg/dL) cholesterol at a local Quest Diagnostics
Low Density Lipoprotein (LDL) cholesterol | Baseline, 3, 6, 9, 12, 18 month
  Fasting venous sample will be obtained for Low Density Lipoprotein (LDL, mg/dL) cholesterol at a local Quest Diagnostics
Fasting venous sample | Baseline, 3, 6, 9, 12, 18 month
  Fasting venous sample will be obtained for triglyceride level (mg/dL) at a local Quest Diagnostics
8-year Diabetes Risk | Baseline, 3, 6, 9, 12, 18 month
  The Framingham Heart Study diabetes risk score will be calculated by combining age, gender, fasting glucose, body mass index, HDL cholesterol and triglyceride levels, blood pressure, and parental history of diabetes. Risk score calculator and regression model are free and used in GLB weight-loss trials
Metabolic Syndrome Severity Score | Baseline, 3, 6, 9, 12, 18 month
  Metabolic Syndrome is a cluster of cardiovascular risk factors that include large waist circumference, high body mass index [BMI]), high blood pressure, high triglycerides, low high density lipoprotein (HDL) cholesterol and high fasting blood sugar (HBA1c). The score is calculated by combining these risk factors into a calculator. Individuals who have ≥3 of these risk factors have metabolic syndrome, placing them at greater risk of developing heart disease and diabetes. Risk scores below 0 indicate a lower degree of metabolic syndrome risk than the average US adult; scores above 0 are associated with greater risk for disease. A score of 1 indicates risk is higher than 84.1% of US adults and a score of 2 is higher than 97.7% of US adults. Z scores are calculated for BMI and waist circumference.
Behavioral Risk Factor Surveillance System (BRFSS) | Baseline, 3, 6, 9, 12, 18 month
  The Behavioral Risk Factor Surveillance System (BRFSS) is a state-based system of health surveys that collects information on health risk behaviors, preventative health practices, and health care access primarily related to chronic disease and injury. Investigators will use the two subscales of Healthy Eating and Physical Activity from the 2017 version of the BRFSS. It consists of 14 items.
Substance Use | Baseline, 12, 18 month
  Substance use will be assessed using a brief survey of tobacco use (cigarettes, chewing tobacco), drug use (illicit or non-prescription drugs), and alcohol use.
Neighborhood Environment Walkability Scale (NEWS) | Baseline, 3, 6, 9, 12, 18 month
  Neighborhood Environment Walkability Scale (NEWS) assesses participants' perception of neighborhood features related to physical activity and grocery shopping, including residential density, land use mix (including both indices of proximity and accessibility), street connectivity, infrastructure for walking/cycling, neighborhood aesthetics, traffic and crime safety, and neighborhood satisfaction. Scores provide insight into environmental barriers faced, are sensitive to behavior change, and can be used as a covariate for weight-loss. Scores are calculated in time to walk to local amenities (minutes) as well as Likert Scale from 1 (strongly disagree) to 4 (strongly agree) to ease of access to local amenities. Higher scores on the Likert Scale and lower scores in time suggest greater walkability.
Quality of Life | Baseline, 3, 6, 9, 12, 18 month
  Quality of life (QOL) will be assessed using the Stroke Impact Scale (SIS), which assesses 8 dimensions of health-related quality of life specific to people post stroke including subscales (using a 5pt Likert scale) assessing strength, memory and thinking, emotion, communication, activities of daily living, mobility, hand function, and participation/role function. Higher scores represent greater quality of life.
Self-Rated Abilities for Health Practice | Baseline, 3, 6, 9, 12, 18 month
  Measure includes 28 items that assess health practices among people with disabilities and yields a total Health Practices Score plus 4 subscale scores regarding Exercise, Nutrition, Health Practices, and Psychological Well Being. Items are rated on a 5-point scale from 0 'not at all' to 4 'completely.' Scores range from 0-28 with higher scores indicating higher exercise self-efficacy.
Social Support for Healthy Eating (SSEH) | Baseline, 3, 6, 9, 12, 18 month
  The Social Support for Healthy Eating (SSEH) scale is a 10-item self-report questionnaire assessing the frequency of support received from others for healthy eating habits over the past 3 months on scale from 1 (none) to 5 (very often). It is comprised of a five-item Encouragement and a five-item Discouragement subscale. Family and friend support is measured separately. Higher scores represent greater support.
Social Support for Physical Activity (SSPA) | Baseline, 3, 6, 9, 12, 18 month
  The Social Support for Physical Activity (SSPA) scale is a 13-item self-report questionnaire assessing the frequency of support received from others for engaging in physical activity over the past 3 months on scale from 1 (none) to 5 (very often). It is comprised of a 10-item Participation and a three-item Rewards and Punishments subscale. Family and friend support is measured separately.
Care Partner Healthy Lifestyle Support Tool | Baseline, 3, 6, 9, 12, 18 month
  The Care Partner Healthy Lifestyle Support Tool was designed by researchers at BSWRI to measure how much care partner support was provided to participants during the healthy lifestyle intervention. Questions use a 4-point Likert Scale from "never" to "always", with higher scores representing higher support.
Telehealth Usability and Satisfaction | 6, 12, 18 month
  The Telehealth Usability and Satisfaction Scale is a validated assessment that measures 5 usability factors of telehealth (usefulness, ease of use, effectiveness, reliability, and satisfaction). 9 items are scored on level of agreement from 1-7, with higher scores indicating greater agreement. All subscales have good to excellent reliability (α=.79-.92).
Exit Survey & Interview | 12 or 18 month
  Participants will be asked to complete Exit Survey and Focus Group at the 12 or 18-month assessment to provide experience in, and satisfaction with, the telehealth Group Lifestyle Balance for people post stroke (tGLB-CVA) intervention and suggestions for improvement. The focus group questions will focus on their experience, barriers and facilitators to behavior change, and engagement in the program

CONTACTS AND LOCATIONS:
Locations (1):
- Baylor Scott & White Research Institute, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: Undecided